CLINICAL TRIAL: NCT03726814
Title: A Safety and Efficacy Study of Human Peripheral Blood Derived Induced EPCs for Cerebral Hemorrhagic Stroke
Brief Title: A Clinical Study of iEPC Intervent Subjects With Cerebral Hemorrhagic Stroke
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Allife Medical Science and Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EPC-BJYY-01
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EPC treatment group (Experimental)
  Interventions: Biological: EPC treatment group

INTERVENTIONS:
Biological: EPC treatment group — Brain injection EPC

SUMMARY:
This is a single centre、single arm、open-label，to investigate the safety and efficacy of EPC transplantation in the brain

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of transplantation EPCs intervent subjests with cerebral hemorrhagic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 18 and ≤ 80 years of age
2. Subjects was confirmed cerebral hemorrhagic stroke, included at least one of risk factors(Hypertension, diabetes, coronary heart disease, high blood lipid), and Satisfied with one of the following conditions:

   A. Significant stenosis (> 50%) of the intracranial and extracranial arteries or their branches due to atherosclerosis, or clinical or imaging manifestations of vascular blockage B. Head imaging (CT or MRI) : cerebral hemispheric infarct lesion diameter of > 1.5cm; Or there were more than 2 discontinuous lesions in the blood supply area of the same intracranial external artery.

   C. Auxiliary examination: color ultrasonography, CTA, MRA or DSA of the blood vessels in the neck confirmed that the intracranial or extracranial stenosis was greater than or equal to 50%；
3. Serum creatinine ≤ 1.5 mg/dl ； Serum ALT/AST）≤2.5×ULN；ALB≥25g/L；
4. Serum creatinine≤ 176.8umol/L（2.0 mg/dl）；
5. Prothrombin time（PT）≤15s，International standardization rates（INR）<1.7；
6. The glucose should be control between 2.8~22.2mmol/L（50~400mg/dl）；
7. Adult patients were willing to use reliable contraceptives (such as condoms) and not to donate sperm throughout the study period and within three months of discharge
8. Subjects and the guardians able to undergo post-physical therapy/rehabilitation

Exclusion Criteria:

1. Non-atherogenic cerebral infarction: cardiogenic embolization, small artery occlusion type IS, other exact etiology IS, and unknown etiology IS
2. Combined with cerebral hemorrhage or previous intracranial external blood history, arteriovenous malformation and aneurysm history, or prone to hemorrhage (platelet count below 100 x 109/L)
3. The vital signs of subjects are not stable
4. Subjects with Class III/IV cardiovascular disability according to the New York Heart Association Classification
5. At rest systolic pressure of 170mmHg or diastolic pressure of 105mmHg, or other indications of uncontrolled hypertension
6. Subjects have one kinds of tumors within 5 years
7. The subject was suffering from neurological or mental illness
8. Subjects had congenital or acquired immune deficiencies, active tuberculosis and other active infections (e.g., pulmonary infection, urinary tract infection, skin infection)
9. alcoholics
10. Receipt of any investigational drug or device within 3 month
11. Active hepatitis B (HBV DNA>1000copy/mL), hepatitis C or HIV infection
12. Subjects who have other conditions that were not appropriate for the group determined by the researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent AE | 1 year
  Defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment